CLINICAL TRIAL: NCT01841385
Title: Influence of Application of the Pilates Method on Pulmonary Function, Thoracic Mobility and Respiratory Muscle Strength
Brief Title: Effects of Pilates on Respiratory Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Eli Maria Pazzianotto Forti, PhD, Universidade Metodista de Piracicaba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pilates2012
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Exercise
Keywords: Exercise; spirometry; muscle strength; physical therapy modalities
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilates Group (Experimental): Sedentary volunteers, but that would begin activities with the Pilates method and evaluated in three months.
  Therapeutic intervention in the Pilates method has two regular weekly sessions for 12 weeks, totaling 24 sessions.
  For the protocol of Pilates exercises, exercises on soil and equipment, with gradual progression of the load.
  Interventions: Other: Pilates method
- Control Group (No Intervention): Sedentary volunteers and remain sedentary and evaluated in three months. The volunteers comprised the control group did not perform any physical activity during the study period.

INTERVENTIONS:
Other: Pilates method — Therapeutic intervention in the Pilates method has two regular weekly sessions for 12 weeks, totaling 24 sessions. For the protocol of Pilates exercises, exercises on soil and equipment, with gradual progression of the load.
  Arms: Pilates Group

SUMMARY:
The aim of this study was to evaluate the influence of a fitness program from the application of Pilates on lung function, thoracoabdominal mobility and respiratory muscle strength in women.

DETAILED DESCRIPTION:
Study in the Cardiorespiratory Physiotherapy laboratory and clinics of Pilates in the region, in which the voluntary of the Pilates group would start the Pilates method.

The study included women with body mass index (BMI) ≤ 29 kg/m2 were not engaged in regular physical activity, or sedentary lifestyle with scores up to eight, according to Baecke et al., non-smoker, non-alcoholic, without any abnormalities of the cardiovascular, respiratory and neuromuscular.

The study excluded women with disabling diseases, pregnancy, postpartum less than a year, inability to understand the tests and exercises proposed or refuse to participate in the study.

The volunteers, aged between 25 and 55 years, were allocated in to two groups:

1. Pilates Group (n = 16): sedentary volunteers, but that would begin activities with the Pilates method and evaluated three months.
2. Control group (n = 13): sedentary volunteers and remain sedentary and evaluated in three months.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≤ 29 kg/m2
* not physically active on a regular basis, ie, sedentary lifestyle with scores up to eight, according to Baecke et al.
* nonsmokers
* non-alcoholic
* without any abnormalities in the cardiovascular, respiratory or neuromuscular

Exclusion Criteria:

* disabling diseases
* gestation
* puerperium there is less than a year
* inability to understand the tests and exercises proposed

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | Three months
  Spirometry was carried out according to the guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS) (2005). Three types of maneuver were used in order to evaluate the lung volumes and flows: Slow Vital Capacity (SVC), Forced Vital Capacity (FVC) and Maximum Voluntary Ventilation (MVV). The maneuvers were carried out until three acceptable and reproducible curves were obtained, not exceeding more than eight attempts. The values extracted from each maneuver were selected according to Pereira (2002), and the predicted values calculated using the equation proposed by Pereira et al. (1992) for Brazilians.
Thoracoabdominal mobility | Three months
  The measurement of thoracoabdominal mobility was performed by using a tape scaled in centimeters. In the standing position, the measurements were made at levels axillary, xiphoid and abdominal, during rest, and at maximal inspiration and maximal expiration. At each level, the measurements were performed three times. It computed the highest value of inspiration and the lowest of expiration. The absolute difference between these values was considered the thoracoabdominal mobility.
Respiratory muscle strength | Three months
  Respiratory muscle strength was assessed by measuring maximal respiratory pressures (MRP) with the use of an analog manometer, with operating range of ± 300 cmH2O.
  The maximal inspiratory pressure (MIP) was measured from a maximal expiration, near the residual volume. The maximal expiratory pressure (MEP) was measured from a maximal inspiration, near total lung capacity. Each inspiratory or expiratory effort was sustained for at least two seconds and was respected the 45 seconds between each maneuver.
  To minimize the learning effect five measurements were performed and the difference between them should be as high as 10%. Was considered for analysis the highest value obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Metodista de Piracicaba (UNIMEP), Piracicaba, São Paulo, Brazil